CLINICAL TRIAL: NCT03867019
Title: The Cardiac Autonomic Control System Response to Vestibular Stimulation in Subjects With and Without BPPV
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Moshe Chaimoff, Dr. Moshe Chaimoff, Otolaryngology specialist, Principal investigator, Clalit Health Services
Other Study IDs: 0179-18-COM1
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Benign Paroxysmal Positional Vertigo; Vertigo; Autonomic Nervous System
Keywords: Benign Paroxysmal Positional Vertigo; BPPV; Vertigo; Autonomic Nervous System; Heart Rate Variability; Vestibulo Sympathetic Response; Vestibulo Sympathetic Reflex
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with BPPV: Patients diagnosed with BPPV, who meet the following criteria:
  1. Main complain of spinning sensation (Vertigo) when changes are made in head position relative to gravity.
  2. Positive Dix-Hallpike / Supine Roll Test, confirmed by presence of nystagmus.
  Interventions: Diagnostic Test: Heart rate variability parameters monitoring
- Subjects without BPPV (Control group): Patients who do not suffer from dizziness / spinning sensation (Vertigo), and do not meet the exclusion criteria in the study.
  Interventions: Diagnostic Test: Heart rate variability parameters monitoring

INTERVENTIONS:
Diagnostic Test: Heart rate variability parameters monitoring — No intervention- only additional monitoring of heart rate, physical tests and filling of questionnaires:
  Heart rate variability parameters monitoring- by wearing a Polar watch (RS800CX).
  Isometric grip test- by using a Jamar Hand Held Dynamometer.
  Questionnaires:
  1. Dizziness Handicap Inventory (DHI) - hebrew version.
  2. Stait-Trait Anxiety Inventory (STAI)
  Other Names: Isometric grip test; Five times sit to stand; Questionnaires

SUMMARY:
The vestibular system in the inner year is an important system in the body which is responsible for balance. In addition, there is evidence that the vestibular system plays a role in maintaining blood pressure while changing body position, such as moving from lying down in bed to sitting. Dysfunction of the vestibular system may affect the ability to maintain blood pressure, therefore the aim of this study is to assess if a specific problem in the vestibular system (Benign Paroxysmal Positional Vertigo- BPPV) may cause changes in the interaction between the vestibular system and the cardiovascular system. We assume that patients with this medical condition (BPPV) will have different heart rate parameters in comparison with healthy patients.

DETAILED DESCRIPTION:
This is a case-control study, that will consist of one routine assessment by a vestibular physiotherapist in an outpatient clinic in Tel Aviv ("Clalit Health Services"). The session will last approximately 90 minutes, and will include 40-60 participants.

Two groups of patients (30-70 years old) will be assigned to this study:

1. Patients with Benign Paroxysmal Positional Vertigo (BPPV).
2. Healthy patients (Control Group).

Both groups will undergo routine physical assessment which is done to diagnose if the patient has BPPV or not. The physical assessment includes quick changes in body and head position.

In addition to the routine physical assessment, heart rate variability parameters will be monitored during the whole session in patients in both groups (using Polar watch RS800CX). Furthermore, all patients will be asked to test their grip strength (using a hand-held dynamometer), moving from sitting to standing 5 times in a row and to fill two questionnaires.

The patients that were diagnosed with BPPV will be treated with the routine vestibular physiotherapy, performed by the same physiotherapist who did the physical assessment.

Statistical analysis of the data will be performed in IBM SPSS Statistics software (version 24), and a statistical significance level of a p-value < 0.05 will be considered significant. Normality distribution will be tested with the Kolmagorov-Smirnov test.

Parametric tests suitable for the analysis of the data in this study are:

1. Paired and unpaired t-tests.
2. Repeated Measures Analysis of Variance (ANOVA).

Non-parametric tests suitable for the analysis of the data in this study are:

1. Mann-Whitney.
2. Wilcoxon.

Spearman coefficient will be used to examine correlations.

ELIGIBILITY:
Inclusion Criteria:

Subjects with BPPV- Patients diagnosed with BPPV, who meet the following criteria:

1. Main complain of spinning sensation (Vertigo) when changes are made in head position relative to gravity (such as when moving from sitting to lying down or rolling in bed, bending over etc.)
2. Positive Dix-Hallpike / Supine Roll Test, confirmed by presence of nystagmus.

Subjects without BPPV (Control group):

Subjects who do not suffer from dizziness / spinning sensation (Vertigo).

Exclusion Criteria:

* Suffering from pain in the day of assessment.
* Postural Hypotension.
* Familial Dysautonomia.
* Diabetic Neuropathy.
* History of Whiplash or Traumatic Brain Injury (TBI) in the last year.
* History of Stroke (CVA), Multiple Sclerosis (MS) or Central Positional Vertigo.
* Coronary Heart Disease (CHD), Cardiac Heart Failure (CHF), Cardiac arrhythmias, Vertebrobasilar Insufficiency (VBI).
* Under treatment of Beta- Blockers.
* Anxiety Disorders.
* Vestibular Migraine, Vestibular Neuritis, Menier's Disease, Perilymphatic Fistula, Superior Canal Dehiscence Syndrome.
* Medical conditions with high risk of subluxation / dislocation of the Atlanto-axial joint.
* Health professionals who are specialized to treat Vestibular disorders (such as Vestibular physiotherapists)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without BPPV will be recruited to the study in an outpatient physiotherapy clinic (community sample), "Clalit Health Services", in Tel Aviv.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability- SDNN | Through study completion, approximately 1 year
  Standard Deviation of the Normal to Normal intervals
Heart Rate Variability- RMSSD | Through study completion, approximately 1 year
  Root Mean Square of the Successive Differences

SECONDARY OUTCOMES:
Dizziness Handicap Inventory | Through study completion, approximately 1 year
  Dizziness Handicap Inventory score from the hebrew version of the questionnaire
Stait- Trait Anxiety Inventory | Through study completion, approximately 1 year
  Stait- Trait Anxiety Inventory score from the hebrew version of the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Chaimoff, Dr., Principal Investigator — Clalit Health Services
Locations (1):
- Horowitz Physiotherapy Clinic, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ▪ Bhattacharyya, N., Gubbels, S. P., Schwartz, S. R., Edlow, J. A., El-Kashlan, H., Fife, T., ... & Seidman, M. D. (2017). Clinical practice guideline: benign paroxysmal positional vertigo (update). Otolaryngology-Head and Neck Surgery, 156(3_suppl), S1-S47. ▪ Carter, J. R., & Ray, C. A. (2008). Sympathetic responses to vestibular activation in humans. American Journal of Physiology-Regulatory, Integrative and Comparative Physiology, 294(3), R681-R688. ▪ Ewing, D. J., & Clarke, B. F. (1982). Diagnosis and management of diabetic autonomic neuropathy. British medical journal (Clinical research ed.), 285(6346), 916. ▪ Ewing, D. J., Irving, J. B., Kerr, F., Wildsmith, J. A. W., & Clarke, B. F. (1974). Cardiovascular responses to sustained handgrip in normal subjects and in patients with diabetes mellitus: a test of autonomic function. Clinical Science, 46(3), 295-306. ▪ Fielder, H., Denholm, S. W., Lyons, R. A., & Fielder, C. P. (1996). Measurement of health status in patients with vertigo. Clinical Otolaryngology, 21(2), 124-126. ▪ Jacob, R. G., & Furman, J. M. (2001). Psychiatric consequences of vestibular dysfunction. Current opinion in Neurology, 14(1), 41-46. ▪ Jáuregui-Renaud, K., Aw, S. T., Todd, M. J., McGarvie, L. A., & Halmagyi, G. M. (2005). Benign paroxysmal positional vertigo can interfere with the cardiac response to head-down tilt. Otology & Neurotology, 26(3), 484-488. ▪ Jáuregui-Renaud, K., Hermosillo, A. G., Gómez, A., Márquez, M. F., Cárdenas, M., & Bronstein, A. M. (2003). Autonomic function interferes in cardiovascular reflexes. Archives of medical research, 34(3), 200-204. ▪ Julian, L. J. (2011). Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis care & research, 63(S11). ▪ Kaplan DM, Friger M, Racover NK, Peleg A, Kraus M, Puterman M. [The Hebrew dizziness handicap inventory]. Harefuah. 2010 Nov;149(11):697-700, 750, 749.Hebrew. PubMed PMID: 21250408 ▪ Khurana, R. K., & Setty, A. (1996). The value of the isometric hand-grip test-studies in various autonomic disorders. Clinical Autonomic Research, 6(4), 211-218. ▪ McCall, A. A., Miller, D. M., & Yates, B. J. (2017). Descending influences on vestibulospinal and vestibulosympathetic reflexes. Frontiers in neurology, 8, 112. ▪ Mutlu, B., & Serbetcioglu, B. (2013). Discussion of the dizziness handicap inventory. Journal of Vestibular Research, 23(6), 271-277. ▪ Nussinovitch, U., Elishkevitz, K. P., Katz, K., Nussinovitch, M., Segev, S., Volovitz, B., & Nussinovitch, N. (2011). Reliability of ultra-short ECG indices for heart rate variability. Annals of Noninvasive Electrocardiology, 16(2), 117-122. ▪ Ray, C. A. (2000). Interaction of the vestibular system and baroreflexes on sympathetic nerve activity in humans. American Journal of Physiology-Heart and Circulatory Physiology, 279(5), H2399-H2404. ▪ Schroeder, E. B., Whitsel, E. A., Evans, G. W., Prineas, R. J., Chambless, L. E., & Heiss, G. (2004). Repeatability of heart rate variability measures. Journal of electrocardiology, 37(3), 163-172. ▪ Sztajzel, J. (2004). Heart rate variability: a noninvasive electrocardiographic method to measure the autonomic nervous system. Swiss medical weekly, 134(35-36), 514-522. ▪ Yates, B. J., Bolton, P. S., & Macefield, V. G. (2014). Vestibulo-sympathetic responses. Comprehensive Physiology, 4(2), 851-887. ▪ Yates, B. J., & Bronstein, A. M. (2005). The effects of vestibular system lesions on autonomic regulation: observations, mechanisms, and clinical implications. Journal of Vestibular Research, 15(3), 119-129.